CLINICAL TRIAL: NCT02112565
Title: A Phase I, Dose-Escalation, Safety and Tolerability Study of COH29 in Patients With Solid Tumors Refractory to Standard Therapy or for Which No Standard Therapy Exists
Brief Title: RNR Inhibitor COH29 in Treating Patients With Solid Tumors That Are Refractory to Standard Therapy or For Which No Standard Therapy Exists
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14023; NCI-2014-00708 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14023 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (RNR inhibitor COH29) (Experimental): Patients receive RNR inhibitor COH29 PO BID on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: RNR inhibitor COH29; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: RNR inhibitor COH29 — Given PO
  Other Names: COH29; ribonucleotide reductase holoenzyme inhibitor COH29
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of RNR Inhibitor City of Hope 29 (COH29) in treating patients with solid tumors that are refractory to standard therapy or for which no standard therapy exists. COH29 may inhibit an enzyme called ribonucleotide reductase and may interfere with the ability of tumor cells to grow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of COH29 (ribonucleotide reductase [RNR] inhibitor COH29) and recommended dose for further phase II testing.

II. To determine the pharmacokinetics of COH29.

SECONDARY OBJECTIVES:

I. To characterize the safety and tolerability of COH29 by assessing toxicities per Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

II. To characterize any clinical activity of COH29 via objective tumor response.

III. To assess pharmacodynamic response of COH29 on ribonucleotide reductase (RR) and poly-adenosine diphosphate-ribose polymerase (PARP) activity in peripheral blood mononuclear cells (PBMCs).

IV. To explore baseline RRM2 tumor protein expression as a potential correlative marker for COH29 response.

V. To explore measurement of plasma cytokeratin 18 (CK18) as a surrogate pharmacodynamic marker of COH29 antitumor activity.

OUTLINE: This is a dose escalation study.

Patients receive RNR inhibitor COH29 orally (PO) twice daily (BID) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have the ability to understand and the willingness to sign a written informed consent
* Life expectancy of greater than 3 months by physician assessment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have histologically or cytologically confirmed (at original diagnosis or subsequent recurrence or progression) solid tumor that is metastatic, unresectable, progressive, or recurrent, and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have measurable or evaluable disease
* Patients must not have received prior chemotherapy or radiation for < 4 weeks prior to start of study treatment
* Patients may be entered if they have received prior radiation therapy involving =< 30% of the bone marrow; any prior radiation therapy must have been administered >= 4 weeks prior to start of study treatment and the patient must be recovered from the acute toxic effects of the treatment prior to start of study treatment
* Patients may be enrolled with a history of treated brain metastases that are clinically stable for >= 4 weeks prior to start of study treatment
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; women of child-bearing age will undergo urine pregnancy testing prior to study enrollment; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Active breast-feeding is also not allowed on study enrollment
* Leukocytes >= 3,000 cells/µL
* Absolute neutrophil count >= 1,500 cells/µL
* Platelets >= 100, 000 cells/µL
* Total bilirubin =< 1.5 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN; AST/ALT =< 5 x ULN if liver metastasis is present
* Serum creatinine =< 1.5 mg/dL or a measured creatinine clearance >= 50 mL/min
* Prothrombin time (PT)/international normalized ratio (INR)/ activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* Negative serum beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only)

Exclusion Criteria:

* Patients may not be receiving any other investigational agents; use of over-the-counter herbal medications will also be excluded
* Patients with uncontrolled undercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients unable or unwilling to swallow pills
* Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease or heart block, or uncontrolled congestive heart failure
* Patients with a history of noninfectious pneumonitis will be excluded during the dose-escalation phase of the trial
* Patients, who in the opinion of the investigator and another independent party, may not be able to adhere to the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of RNR inhibitor COH29, defined as the dose level with no more than 1 dose limiting toxicity (DLT) in the first 6 patients at a dose level below a dose level with DLT in 2 of 6 patients, graded according to CTCAE version 4.0 | Day 28

SECONDARY OUTCOMES:
Changes in plasma biomarker expression levels | Baseline to up to 30 days after completion of study treatment
  Descriptive statistics and graphical displays will be used to summarize levels of plasma CK18, dNTP pools, gamma-H2AX, and PAR expression at each time point and evaluate changes between pre- and post-treatment measurements. A paired t-test will be used to determine if there is a statistically significant change.
Pharmacokinetics of RNR inhibitor COH29 | Pre-dose and 15 minutes, 30 minutes, 1, 2 , 3, 4, 6, 8, 24, and 168 hours post the day 1, course 1 dose
  COH29 levels in plasma will be quantitated using a validated High Performance Liquid Chromatography (HPLC) tandem mass spectrometry (LC-MS/MS) method. Summary statistics of the pharmacokinetic parameters for the population will be derived from the parameters obtained in individual patients.
Toxicities according to the National Cancer Institute (NCI) CTCAE v 4.0 | Up to 30 days after completion of study treatment
  Toxicities will be tabulated by type and grade.
Response rate | Up to 30 days after completion of study treatment
  Response rate will be estimated in the overall population and 95% exact confidence intervals will be estimated.
RR protein levels as assessed by automated quantitative analysis (AQUA) | Baseline
  Will be summarized descriptively using means, median, standard deviation and range.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States